CLINICAL TRIAL: NCT00449670
Title: Assess the Consistency of the Immunogenicity of a GlaxoSmithKline Biologicals' Pandemic Influenza Vaccine (GSK1562902A) in Adults Aged Between 18 and 60 Years
Brief Title: Assess Consistency of Immunogenicity of GlaxoSmithKline Biologicals' Pandemic Influenza Vaccine (GSK1562902A) in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109630; 109873 (Other: GSK)
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Influenza; Influenza Vaccines
Keywords: Influenza; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- H5N1 Adjuvanted Group (Experimental): Subjects received 2 doses of H5N1 adjuvanted split virus vaccine (lot 1, 2, 3 or 4) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 during Primary Phase. A subset of these subjects (Boosted sub-cohort) received a single dose of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 during Booster Phase. The remaining subjects (Non-Boosted sub-cohort) received a single booster dose at Month 12 or 36 after initial priming in study 111443 (NCT00652743).
  Interventions: Biological: H5N1 adjuvanted split virus vaccine (A/Vietnam/1194/2004 strain); Biological: H5N1 adjuvanted split virus vaccine (A/Indonesia/05/2005 strain)
- H5N1 Un-adjuvanted Group (Active Comparator): Subjects received 2 doses of a H5N1 non-adjuvanted split virus vaccine containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 and two booster doses of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 and Month 6 + 21 days.
  Interventions: Biological: H5N1 non-adjuvanted split virus vaccine (A/Vietnam/1194/2004 strain); Biological: H5N1 adjuvanted split virus vaccine (A/Indonesia/05/2005 strain)

INTERVENTIONS:
Biological: H5N1 adjuvanted split virus vaccine (A/Vietnam/1194/2004 strain) — Two doses of the GSK1562902A adjuvanted split virus vaccine, administered intramuscularly into the deltoid region of the non-dominant arm at Day 0 and Day 21.
  Arms: H5N1 Adjuvanted Group
Biological: H5N1 non-adjuvanted split virus vaccine (A/Vietnam/1194/2004 strain) — Two doses of the GSK1562902A non-adjuvanted split virus vaccine, administered intramuscularly into the deltoid region of the non-dominant arm at Day 0 and Day 21.
  Arms: H5N1 Un-adjuvanted Group
Biological: H5N1 adjuvanted split virus vaccine (A/Indonesia/05/2005 strain) — Booster administration at Month 6 (and a second booster dose 21 days later for the un-adjuvanted group only) with an adjuvanted split virus pandemic influenza candidate vaccine containing the strain A/Indonesia/5/2005.

SUMMARY:
The present study is designed to assess the lot-to-lot consistency of the immunogenicity of a GlaxoSmithKline Biologicals' pandemic influenza candidate vaccine (GSK1562902A) in adults aged between 18 and 60 years.

DETAILED DESCRIPTION:
The protocol posting has been updated to reflect changes due to an amendment to the protocol (addition of an exclusion criterion). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* A male or female between, and including, 18 and 60 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Administration of any licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol during the following periods: from Day 0 up to Day 51, 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to Month 6; from Month 6 up to Month 6 + 30 days (or Month 6 + 51 days for the control groups).
* Previous vaccination with a pandemic candidate vaccine or a vaccine containing the same adjuvant as the study vaccine.
* Previous proven contact with H5N1 wild type virus (i.e. contact with an individual with laboratory-confirmed H5N1 infection, or contact with an animal (e.g. poultry) which died as a result of H5N1 infection).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first administration of the candidate vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, or autoimmune diseases such as Guillain Barre Syndrome, based on medical history and physical examination (no laboratory testing required).
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first administration of the candidate vaccine or during the study.
* Lactating women.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1206 (Actual)
Dates: Start 2007-03-24 (Actual); Primary Completion 2007-07-12 (Actual); Study Completion 2008-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Hong Kong, Hong Kong
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chu DW, Hwang SJ, Lim FS, Oh HM, Thongcharoen P, Yang PC, Bock HL, Drame M, Gillard P, Hutagalung Y, Tang H, Teoh YL, Ballou RW; H5N1 Flu Study Group for Hong Kong, Singapore, Taiwan and Thailand. Immunogenicity and tolerability of an AS03(A)-adjuvanted prepandemic influenza vaccine: a phase III study in a large population of Asian adults. Vaccine. 2009 Dec 9;27(52):7428-35. doi: 10.1016/j.vaccine.2009.07.102. Epub 2009 Aug 13. PMID 19683087
- [Background] Chu DW, Kwong AS, Tsui WW, Wang JH, Ngai CK, Wan PK, Ong G, Tang HW, Roman F, Dram M, Bock HL. Cross-clade immunogenicity and safety of an AS03A-adjuvanted prepandemic H5N1 influenza vaccine in Hong Kong. Hong Kong Med J. 2011 Feb;17(1):39-46. PMID 21282825
- [Background] Hwang SJ, Chang SC, Yu CJ, Chan YJ, Chen TJ, Hsieh SL, Lai HY, Lin MH, Liu JY, Ong G, Roman F, Drame M, Bock HL, Yang PC. Immunogenicity and safety of an AS03(A)-adjuvanted H5N1 influenza vaccine in a Taiwanese population. J Formos Med Assoc. 2011 Dec;110(12):780-6. doi: 10.1016/j.jfma.2011.11.009. Epub 2011 Dec 23. PMID 22248833
- [Background] Thongcharoen P, Auewarakul P, Hutagalung Y, Ong G, Gillard P, Drame M, Bock HL. Cross-clade immunogenicity and antigen-sparing with an AS03(A)-adjuvanted prepandemic influenza vaccine in a Thai population. J Med Assoc Thai. 2011 Aug;94(8):916-26. PMID 21863672
- [Background] Gillard P, Chu DW, Hwang SJ, Yang PC, Thongcharoen P, Lim FS, Drame M, Walravens K, Roman F. Long-term booster schedules with AS03A-adjuvanted heterologous H5N1 vaccines induces rapid and broad immune responses in Asian adults. BMC Infect Dis. 2014 Mar 15;14:142. doi: 10.1186/1471-2334-14-142. PMID 24628789
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109630 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- H5N1 Un-adjuvanted Group: Subjects received 2 doses of a H5N1 non-adjuvanted split virus vaccine(lot 1 or 2) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 and two booster doses of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 and Month 6 + 21 days.
Period: Primary Phase (Study no.109630)
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Started | 961 | 245
Completed | 947 | 243
Not Completed | 14 | 2
Not completed — Serious Adverse Event | 1 | 0
Not completed — Non-serious adverse event | 4 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 5 | 1
Period: Booster Phase (Study no.109873)
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Started | 265 | 236
Completed | 265 | 233
Not Completed | 0 | 3
Not completed — Migrated/moved from study area | 0 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group | Total
Number analyzed (Participants) | 961 | 245 | 1206
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (9.82) | 32.95 (9.18) | 33.59 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 495 | 122 | 617
  Male | 466 | 123 | 589
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian - Central/ South Asian Heritage | 16 | 6 | 22
  Race: Asian - East Asian Heritage | 589 | 145 | 734
  Race: Asian - South East Asian Heritage | 355 | 93 | 448
  Race: White - Arabic / North African Heritage | 0 | 1 | 1
  Race: White - Caucasian / European Heritage | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1). The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: Before vaccination (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for Immunogenicity, which included all vaccinated and eligible subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- H5N1 Adjuvanted Group - Lot 1: Subjects received 2 doses of H5N1 adjuvanted split virus vaccine (lot 1) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 during Primary Phase. A subset of these subjects (Boosted sub-cohort) received a single dose of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 during Booster Phase. The remaining subjects (Non-Boosted sub-cohort) received a single booster dose at Month 12 or 36 after initial priming in study 111443 (NCT00652743).
- H5N1 Adjuvanted Group - Lot 2: Subjects received 2 doses of H5N1 adjuvanted split virus vaccine (lot 2) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 during Primary Phase. A subset of these subjects (Boosted sub-cohort) received a single dose of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 during Booster Phase. The remaining subjects (Non-Boosted sub-cohort) received a single booster dose at Month 12 or 36 after initial priming in study 111443 (NCT00652743).
- H5N1 Adjuvanted Group - Lot 3: Subjects received 2 doses of H5N1 adjuvanted split virus vaccine (lot 3) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 during Primary Phase. A subset of these subjects (Boosted sub-cohort) received a single dose of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 during Booster Phase. The remaining subjects (Non-Boosted sub-cohort) received a single booster dose at Month 12 or 36 after initial priming in study 111443 (NCT00652743).
- H5N1 Adjuvanted Group - Lot 4: Subjects received 2 doses of H5N1 adjuvanted split virus vaccine (lot 4) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 during Primary Phase. A subset of these subjects (Boosted sub-cohort) received a single dose of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 during Booster Phase. The remaining subjects (Non-Boosted sub-cohort) received a single booster dose at Month 12 or 36 after initial priming in study 111443 (NCT00652743).
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 233 | 235 | 231 | 234 | 236
Titers
  A/Vietnam/1194/2004 | 5.6 [5.3 to 5.9] | 5.5 [5.2 to 5.8] | 5.6 [5.2 to 5.9] | 5.4 [5.2 to 5.7] | 5.6 [5.3 to 5.9]
  A/Indonesia/5/2005 | 5.1 [5 to 5.2] | 5 [5 to 5.1] | 5 [5 to 5.1] | 5.1 [5 to 5.1] | 5.0 [5.0 to 5.1]

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: Within 21 days following 2-dose primary vaccination (at Day 42)
Population: Analysis was performed on subjects from H5N1 Adjuvanted Lot Groups, included in the ATP cohort for immunogenicity, for lot-to-lot consistency of the immune response elicited by four compositions of GSK Biological's pandemic influenza candidate vaccine. Analysis was also performed on the subjects from the H5N1 unadjuvanted group
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
Titers
  A/Vietnam/1194/2004 | 192.7 [164.2 to 226.2] | 235.2 [203.1 to 272.5] | 225.6 [193.5 to 263] | 226.3 [194 to 264] | 7.5 [6.7 to 8.3]
  A/Indonesia/5/2005 | 24.3 [20.4 to 29] | 27.9 [23.4 to 33.3] | 25.5 [21.2 to 30.7] | 22.4 [18.6 to 27] | 5.2 [5.0 to 5.4]
Statistical Analysis 1: Comparison: H5N1 Adjuvanted Group - Lot 1 vs H5N1 Adjuvanted Group - Lot 2; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 1 and Lot 2); Test type: Equivalence — The lot-to-lot consistency 21 days after Dose 2 was demonstrated if, for all pairs of lots, the two-sided 95% CIs for the ratio of A/Vietnam/1194/2004 HI antibody GMT was within the [0.5 ; 2] clinical limit interval; ANCOVA; Adjusted GMT ratio = 0.81, 95% CI [0.66 to 1.01]
Statistical Analysis 2: Comparison: H5N1 Adjuvanted Group - Lot 1 vs H5N1 Adjuvanted Group - Lot 3; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 1 and Lot 3); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT ratio = 0.85, 95% CI 2-sided [0.69 to 1.06]
Statistical Analysis 3: Comparison: H5N1 Adjuvanted Group - Lot 1 vs H5N1 Adjuvanted Group - Lot 4; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 1 and Lot 4); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT ratio = 0.85, 95% CI 2-sided [0.68 to 1.05]
Statistical Analysis 4: Comparison: H5N1 Adjuvanted Group - Lot 2 vs H5N1 Adjuvanted Group - Lot 3; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 2 and Lot 3); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT ratio = 1.05, 95% CI 2-sided [0.85 to 1.3]
Statistical Analysis 5: Comparison: H5N1 Adjuvanted Group - Lot 2 vs H5N1 Adjuvanted Group - Lot 4; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 2 and Lot 4); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT ratio = 1.04, 95% CI 2-sided [0.84 to 1.29]
Statistical Analysis 6: Comparison: H5N1 Adjuvanted Group - Lot 3 vs H5N1 Adjuvanted Group - Lot 4; Demonstration of the consistency of the immune response (in terms of geometric mean titer [GMT] ratio for anti-hemagglutinin (anti-HA) antibody response against the A/Vietnam/1194/2004 strain 21 days after the second vaccination) elicited by two compositions of H5N1 adjuvanted vaccine (Lot 3 and Lot 4); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMT ratio = 0.99, 95% CI 2-sided [0.8 to 1.23]

3. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: Within 21 days following the first primary vaccination dose (Day 21)
Population: The analysis was performed on the According-to-Protocol cohort for Immunogenicity, which included all vaccinated and eligible subjects for whom data concerning immunogenicity outcome measures were available, and for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
Titers
  A/Vietnam/1194/2004 | 21.8 [18.1 to 26.2] | 25.1 [20.7 to 30.5] | 24 [19.6 to 29.3] | 20.5 [17 to 24.6] | 6.7 [6.0 to 7.4]
  A/Indonesia/5/2005 | 6.3 [5.7 to 6.8] | 5.9 [5.6 to 6.3] | 5.9 [5.5 to 6.4] | 5.1 [5 to 5.1] | 5.2 [5.0 to 5.3]

4. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: Before booster vaccination at Month 6 (M6) and following booster vaccination at Month 6+21 days (M6+21D) and at Month 6+42 days (M6+42D)
Population: The analysis was performed on the Booster According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who received a booster dose at Month 6 for whom immunogenicity data for the considered assay and timepoint were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 256 | 229
Titers
  A/Vietnam/1194/2004, M6 | 19.1 [16.5 to 22.2] | 5.8 [5.4 to 6.2]
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 256 | 228
  A/Vietnam/1194/2004, M6+21D | 397.4 [342.5 to 461.0] | 30.1 [24.9 to 36.3]
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 0 | 228
  A/Vietnam/1194/2004, M6+42D |  | 76.3 [64.1 to 90.8]
  A/Indonesia/5/2005, M6 | 6.4 [6 to 6.9] | 5.1 [5 to 5.1]
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 256 | 228
  A/Indonesia/5/2005, M6+21D | 321.3 [274.3 to 376.2] | 24.8 [20.5 to 30.0]
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 0 | 228
  A/Indonesia/5/2005, M6+42D |  | 96.3 [80.6 to 115.1]

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: Before booster vaccination at Month 6 (M6) and following booster vaccination at Month 6+21 days (M6+21D) and at Month 6+42 days (M6+42D) and at Month 12 (M12)
Population: The analysis was performed on the Booster ATP cohort for persistence, which included all evaluable subjects who received a booster dose at Month 6, who complied with the protocol during the entire study period and for whom immunogenicity data for the considered assay and timepoint were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 251 | 224
Titers
  A/Vietnam/1194/2004, M6 | 19.4 [16.6 to 22.5] | 5.8 [5.4 to 6.2]
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 251 | 223
  A/Vietnam/1194/2004, M6+21D | 395.3 [339.8 to 459.7] | 31.0 [25.6 to 37.5]
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 0 | 223
  A/Vietnam/1194/2004, M6+42D |  | 78 [65.5 to 92.9]
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 228 | 209
  A/Vietnam/1194/2004, M12 | 76.1 [62.5 to 92.7] | 14.3 [12.2 to 16.8]
  A/Indonesia/5/2005, M6 | 6.5 [6 to 6.9] | 5.1 [5 to 5.1]
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 251 | 223
  A/Indonesia/5/2005, M6+21D | 319.1 [271.7 to 374.7] | 25.5 [21 to 30.9]
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 0 | 223
  A/Indonesia/5/2005, M6+42D |  | 98.5 [82.3 to 117.9]
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 228 | 209
  A/Indonesia/5/2005, M12 | 46.9 [38.3 to 57.4] | 14.6 [12.5 to 17.1]

6. Secondary Outcome: Titers for Serum Neutralizing (SN) Antibodies Against 2 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1). The reference seropositivity cut-off value was ≥ 1:28.
Time Frame: Before vaccination at Day 0 (D0) and within 21 days following 2-dose primary vaccination at Day 42 (D42)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 68 | 74 | 69 | 69 | 71
Titers
  A/Vietnam/1194/2004, D0: number analyzed (Participants) | 68 | 74 | 69 | 68 | 71
  A/Vietnam/1194/2004, D0 | 17.8 [15.4 to 20.5] | 17.8 [15.7 to 20.2] | 18 [15.7 to 20.8] | 16.6 [15.3 to 18.1] | 17.7 [15.4 to 20.4]
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 67 | 73 | 69 | 68 | 71
  A/Vietnam/1194/2004, D42 | 274.4 [232.7 to 323.5] | 330.6 [281.4 to 388.4] | 283.1 [234.2 to 342.3] | 350.4 [293.9 to 417.8] | 29.0 [23.4 to 35.9]
  A/Indonesia/5/2005, D0: number analyzed (Participants) | 68 | 73 | 69 | 69 | 71
  A/Indonesia/5/2005, D0 | 14.6 [14 to 15.3] | 14.8 [14 to 15.7] | 15.3 [13.7 to 17.2] | 14.7 [13.9 to 15.5] | 15.6 [14.4 to 16.7]
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 68 | 73 | 69 | 69 | 71
  A/Indonesia/5/2005, D42 | 74.3 [61.9 to 89.3] | 100.0 [86 to 116.5] | 80.4 [66.7 to 96.9] | 82.1 [69.8 to 96.5] | 16.2 [14.8 to 17.8]

7. Secondary Outcome: Titers for Serum Neutralization (SN) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 184 | 47
Titers
  A/Vietnam/1194/2004, M6 | 170.5 [154.6 to 188.0] | 29.4 [23 to 37.6]
  A/Vietnam/1194/2004, M6+21D | 1660.1 [1435.9 to 1919.4] | 248.1 [187 to 329]
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 0 | 45
  A/Vietnam/1194/2004, M6+42D |  | 447.1 [331.9 to 602.1]
  A/Indonesia/5/2005, M6 | 183.6 [167 to 201.8] | 30.3 [22.8 to 40.1]
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 183 | 47
  A/Indonesia/5/2005, M6+21D | 2917.5 [2490.8 to 3417.3] | 451.9 [357.5 to 571.3]
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 0 | 47
  A/Indonesia/5/2005, M6+42D |  | 1075.8 [834.7 to 1386.6]

8. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease in Adults Who Had Not Received the Booster Dose at Month 6
Description: as for outcome 1
Time Frame: At Day 0, at Day 21, at Day 42, at Month 6 and at Month 12
Population: The analysis was performed on the ATP cohort for persistence, which included all evaluable subjects who did not receive a booster dose at Month 6 (Non-Boosted sub-cohort), who complied with the protocol during the entire study period and for whom immunogenicity data for the considered assay and timepoint were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 665
Titers
  A/Vietnam/1194/2004, D0: number analyzed (Participants) | 663
  A/Vietnam/1194/2004, D0 | 5.6 [5.4 to 5.7]
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 661
  A/Vietnam/1194/2004, D21 | 23.3 [20.8 to 26.1]
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 659
  A/Vietnam/1194/2004, D42 | 215.7 [197.4 to 235.7]
  A/Vietnam/1194/2004, M6 | 18.5 [17 to 20.3]
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 559
  A/Vietnam/1194/2004, M12 | 11.4 [10.4 to 12.5]
  A/Indonesia/5/2005, D0: number analyzed (Participants) | 663
  A/Indonesia/5/2005, D0 | 5.1 [5 to 5.1]
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 661
  A/Indonesia/5/2005, D21 | 6.1 [5.8 to 6.3]
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 659
  A/Indonesia/5/2005, D42 | 24.8 [22.3 to 27.5]
  A/Indonesia/5/2005, M6 | 6.3 [6 to 6.5]
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 559
  A/Indonesia/5/2005, M12 | 6.2 [5.9 to 6.5]

9. Secondary Outcome: Titers for Serum Neutralization (SN) Antibodies Against 2 Strains of Influenza Disease in Adults Who Had Not Received the Booster Dose at Month 6
Description: as for outcome 1
Time Frame: At Month 12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 166
Titers
  A/Vietnam/1194/2004 | 215.5 [191.4 to 242.7]
  A/Indonesia/5/2005 | 57.9 [50.5 to 66.4]

10. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against 2 Strains of Influenza Disease
Description: Seroconversion was defined as: for initially seronegative subjects, antibody titer greater than or equal to ≥ 1:40 after vaccination; and for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At Day 21 (D21) and at Day 42 (D42)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 231 | 233 | 229 | 233 | 234
Participants
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Vietnam/1194/2004, D21 | 97 | 103 | 97 | 96 | 8
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Vietnam/1194/2004, D42 | 213 | 220 | 214 | 219 | 13
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Indonesia/5/2005, D21 | 9 | 4 | 5 | 6 | 0
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Indonesia/5/2005, D42 | 108 | 128 | 118 | 110 | 1

11. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 10
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 254 | 228
Participants
  A/Vietnam/1194/2004, M6 | 96 | 2
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 254 | 227
  A/Vietnam/1194/2004, M6+21D | 244 | 110
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 254 | 227
  A/Vietnam/1194/2004, M6+42D | 0 | 174
  A/Indonesia/5/2005, M6 | 9 | 0
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 254 | 227
  A/Indonesia/5/2005, M6+21D | 241 | 105
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 254 | 227
  A/Indonesia/5/2005, M6+42D | 0 | 188

12. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against 2 Strains of Influenza Disease for Adults Who Received the Booster Dose at Month 6 - Booster Phase
Description: as for outcome 10
Time Frame: Following booster vaccination at Month 6 +21 days (M6+21D) and Month 6 +42 days (M6+42D)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 256 | 228
Participants
  A/Vietnam/1194/2004, M6+21D | 233 | 112
  A/Vietnam/1194/2004, M6+42D | 0 | 173
  A/Indonesia/5/2005, M6+21D | 241 | 106
  A/Indonesia/5/2005, M6+42D | 0 | 189

13. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against 2 Strains of Influenza Disease for Adults Who Received the Booster Dose at Month 6 - Booster Phase
Description: as for outcome 10
Time Frame: At Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 228 | 209
Participants
  A/Vietnam/1194/2004 | 93 | 57
  A/Indonesia/5/2005 | 140 | 67

14. Secondary Outcome: Number of Seroconverted Subjects for Neutralizing Antibodies Against 2 Strains of Influenza Disease
Description: Seroconversion was defined as: antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: Within 21 days following 2-dose primary vaccination at Day 42
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 68 | 73 | 69 | 69 | 71
Participants
  A/Vietnam/1194/2004: number analyzed (Participants) | 67 | 73 | 69 | 68 | 71
  A/Vietnam/1194/2004 | 64 | 70 | 64 | 68 | 23
  A/Indonesia/5/2005 | 61 | 70 | 61 | 63 | 4

15. Secondary Outcome: Number of Seroconverted Subjects for Neutralizing Antibodies Against 2 Strains of Influenza Disease - Booster Phase
Description: Seroconversion was defined as: for initially seronegative subjects, antibody titer ≥ 1:56 after vaccination; and for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer.
Time Frame: Following booster vaccination at Month 6+21 days (M6+21D) and at Month 6+42 days (M6+42D)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 184 | 47
Participants
  A/Vietnam/1194/2004, M6+21D | 140 | 36
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 184 | 45
  A/Vietnam/1194/2004, M6+42D | 0 | 41
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 183 | 47
  A/Indonesia/5/2005, M6+21D | 165 | 41
  A/Indonesia/5/2005, M6+42D | 0 | 45

16. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against 2 Strains of Influenza Disease for Adults Who Have Not Received Booster at Month 6
Description: Seroconversion defined as: for initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; and for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-booster antibody titer.
Time Frame: At Day 21, Day 42, Month 6 and Month 12 following primary vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 663
Participants
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 661
  A/Vietnam/1194/2004, D21 | 293
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 659
  A/Vietnam/1194/2004, D42 | 620
  A/Vietnam/1194/2004, M6 | 228
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 558
  A/Vietnam/1194/2004, M12 | 108
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 661
  A/Indonesia/5/2005, D21 | 18
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 659
  A/Indonesia/5/2005, D42 | 328
  A/Indonesia/5/2005, M6 | 11
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 558
  A/Indonesia/5/2005, M12 | 25

17. Secondary Outcome: Number of Seroconverted Subjects for Neutralizing Antibodies Against 2 Strains of Influenza Disease for Subjects Not Boosted at Month 6
Description: as for outcome 15
Time Frame: At Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 23
Participants
  A/Vietnam/1194/2004, M12 | 20
  A/Indonesia/5/2005, M12 | 15

18. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: At day 21 and Day 42
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 231 | 233 | 229 | 233 | 234
Fold change
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Vietnam/1194/2004, D21 | 3.9 [3.3 to 4.6] | 4.6 [3.8 to 5.6] | 4.3 [3.5 to 5.2] | 3.8 [3.2 to 4.5] | 1.2 [1.1 to 1.3]
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Vietnam/1194/2004, D42 | 34.4 [29.2 to 40.5] | 43.2 [37 to 50.5] | 40.5 [34.6 to 47.5] | 41.6 [35.6 to 48.5] | 1.3 [1.2 to 1.5]
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Indonesia/5/2005, D21 | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3] | 1.0 [1.0 to 1.0]
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Indonesia/5/2005, D42 | 4.8 [4 to 5.7] | 5.6 [4.6 to 6.6] | 5.1 [4.2 to 6.1] | 4.4 [3.7 to 5.3] | 1.0 [1.0 to 1.1]

19. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 18
Time Frame: Before booster vaccination at Month 6 (M6) and within 21 days following each booster dose: At Month 6 + 21 days (M6+21D) and, for H5N1 Un-adjuvanted Group only, at Month 6 + 42 days (M6+42D)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 254 | 228
Fold change
  A/Vietnam/1194/2004, M6 | 3.6 [3.1 to 4.1] | 1 [1 to 1.1]
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 254 | 227
  A/Vietnam/1194/2004, M6+21D | 74 [63.1 to 86.7] | 5.3 [4.4 to 6.4]
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 0 | 227
  A/Vietnam/1194/2004, M6+42D |  | 13.4 [11.2 to 16.0]
  A/Indonesia/5/2005, M6 | 1.3 [1.2 to 1.4] | 1 [1 to 1]
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 254 | 227
  A/Indonesia/5/2005, M6+21D | 63.8 [54.4 to 74.9] | 4.9 [4 to 5.9]
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 0 | 227
  A/Indonesia/5/2005, M6+42D |  | 18.9 [15.8 to 22.6]

20. Secondary Outcome: Booster Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 18
Time Frame: Within 21 days following each booster dose: At Month 6 + 21 days (M6+21D) and, for H5N1 Un-adjuvanted Group only, at Month 6 + 42 days (M6+42D)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 256 | 228
Fold change
  A/Vietnam/1194/2004, M6+21D | 20.8 [17.3 to 24.9] | 5.2 [4.3 to 6.2]
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 0 | 228
  A/Vietnam/1194/2004, M6+42D |  | 13.2 [11.1 to 15.8]
  A/Indonesia/5/2005, M6+21D | 50 [42.5 to 58.8] | 4.9 [4.1 to 5.9]
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 0 | 228
  A/Indonesia/5/2005, M6+42D |  | 19 [15.9 to 22.7]

21. Secondary Outcome: Booster Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 18
Time Frame: At Month 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 228 | 209
Fold change
  A/Vietnam/1194/2004 | 3.7 [3.1 to 4.5] | 2.5 [2.1 to 2.9]
  A/Indonesia/5/2005 | 7.2 [5.9 to 8.8] | 2.9 [2.5 to 3.4]

22. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease for Subjects Not Boosted at Month 6
Description: as for outcome 18
Time Frame: At Day 21, at Day 42, at Month 6 and at Month 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 663
Fold change
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 661
  A/Vietnam/1194/2004, D21 | 4.2 [3.8 to 4.7]
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 659
  A/Vietnam/1194/2004, D42 | 38.8 [35.4 to 42.5]
  A/Vietnam/1194/2004, M6 | 3.3 [3.1 to 3.6]
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 558
  A/Vietnam/1194/2004, M12 | 2 [1.9 to 2.2]
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 661
  A/Indonesia/5/2005, D21 | 1.2 [1.2 to 1.3]
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 659
  A/Indonesia/5/2005, D42 | 4.9 [4.4 to 5.4]
  A/Indonesia/5/2005, M6 | 1.2 [1.2 to 1.3]
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 558
  A/Indonesia/5/2005, M12 | 1.2 [1.2 to 1.3]

23. Secondary Outcome: Number of Subjects Seroprotected Against 2 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 2 flu strains assessed were A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1).
Time Frame: Before primary vaccination at Day 0 and within 21 days following each primary vaccination dose at Day 21 and at Day 42.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 233 | 235 | 231 | 234 | 236
Participants
  A/Vietnam/1194/2004, PRE | 4 | 3 | 5 | 3 | 5
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Vietnam/1194/2004, D21 | 102 | 108 | 102 | 100 | 16
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Vietnam/1194/2004, D42 | 213 | 223 | 215 | 220 | 24
  A/Indonesia/5/2005, PRE | 1 | 0 | 0 | 0 | 0
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 231 | 233 | 228 | 233 | 234
  A/Indonesia/5/2005, D21 | 10 | 4 | 6 | 7 | 0
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 229 | 233 | 229 | 233 | 234
  A/Indonesia/5/2005, D42 | 108 | 128 | 118 | 110 | 1

24. Secondary Outcome: Number of Subjects Seroprotected Against 2 Strains of Influenza Disease
Description: as for outcome 23
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 256 | 229
Participants
  A/Vietnam/1194/2004, M6 | 103 | 4
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 256 | 228
  A/Vietnam/1194/2004, M6+21D | 247 | 121
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 256 | 228
  A/Vietnam/1194/2004, M6+42D | 0 | 180
  A/Indonesia/5/2005, M6 | 9 | 0
  RA/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 256 | 228
  RA/Indonesia/5/2005, M6+21D | 243 | 106
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 256 | 228
  A/Indonesia/5/2005, M6+42D | 0 | 189

25. Secondary Outcome: Number of Seroprotected Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 23
Time Frame: Before booster vaccination at Month 6 (M6) and following booster vaccination at Month 6+21 days (M6+21D), at Month 6+42 days (M6+42D) and at Month 12 (M12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 251 | 224
Participants
  A/Vietnam/1194/2004, M6 | 103 | 4
  A/Vietnam/1194/2004, M6+21D: number analyzed (Participants) | 251 | 223
  A/Vietnam/1194/2004, M6+21D | 242 | 120
  A/Vietnam/1194/2004, M6+42D: number analyzed (Participants) | 251 | 223
  A/Vietnam/1194/2004, M6+42D | 0 | 177
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 228 | 209
  A/Vietnam/1194/2004, M12 | 178 | 65
  A/Indonesia/5/2005, M6 | 9 | 0
  A/Indonesia/5/2005, M6+21D: number analyzed (Participants) | 251 | 223
  A/Indonesia/5/2005, M6+21D | 238 | 105
  A/Indonesia/5/2005, M6+42D: number analyzed (Participants) | 251 | 223
  A/Indonesia/5/2005, M6+42D | 0 | 186
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 228 | 209
  A/Indonesia/5/2005, M12 | 151 | 67

26. Secondary Outcome: Number of Subjects Seroprotected Against 2 Strains of Influenza Disease for Subjects Not Boosted at Month 6
Description: as for outcome 23
Time Frame: At Day 0, Day 21, Day 42, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 665
Participants
  A/Vietnam/1194/2004, PRE: number analyzed (Participants) | 663
  A/Vietnam/1194/2004, PRE | 11
  A/Vietnam/1194/2004, D21: number analyzed (Participants) | 661
  A/Vietnam/1194/2004, D21 | 307
  A/Vietnam/1194/2004, D42: number analyzed (Participants) | 659
  A/Vietnam/1194/2004, D42 | 623
  A/Vietnam/1194/2004, M6 | 247
  A/Vietnam/1194/2004, M12: number analyzed (Participants) | 559
  A/Vietnam/1194/2004, M12 | 131
  A/Indonesia/5/2005, PRE: number analyzed (Participants) | 663
  A/Indonesia/5/2005, PRE | 1
  A/Indonesia/5/2005, D21: number analyzed (Participants) | 661
  A/Indonesia/5/2005, D21 | 21
  A/Indonesia/5/2005, D42: number analyzed (Participants) | 659
  A/Indonesia/5/2005, D42 | 328
  A/Indonesia/5/2005, M6 | 13
  A/Indonesia/5/2005, M12: number analyzed (Participants) | 559
  A/Indonesia/5/2005, M12 | 26

27. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 4+ (CD4+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation
Description: The analyzed cytokines were CD 40 Ligand (CD40L), Interleukin 2 (IL-2), Tumor Necrosis Factor-α (TNF-α) and Interferon-γ (IFN-γ). The stimulating antigen used was A/Vietnam/1194/2004.
Time Frame: Within 21 days of each primary vaccine dose: at Day 21 and at Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-cells per million T-cells
Groups:
- H5N1 Un-Adjuvanted Group - Lot 1: Subjects received 2 doses of a H5N1 non-adjuvanted split virus vaccine (lot 1) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 and two booster doses of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 and Month 6 + 21 days.
- H5N1 Un-Adjuvanted Group - Lot 2: Subjects received 2 doses of a H5N1 non-adjuvanted split virus vaccine (lot 2) containing A/Vietnam/1194/2004 strain at Day 0 and Day 21 and two booster doses of heterologous H5N1 adjuvanted vaccine containing A/Indonesia/05/2005 strain at Month 6 and Month 6 + 21 days.
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-Adjuvanted Group - Lot 1 | H5N1 Un-Adjuvanted Group - Lot 2
Number analyzed (Participants) | 6 | 7 | 6 | 4 | 4 | 5
T-cells per million T-cells
  A/Vietnam/1194/2004, min. 2 cytokines, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min. 2 cytokines, D21 | 2602.17 (1369.03) | 5627.00 (3064.90) | 3632.00 (1884.23) | 4060.75 (1566.75) | 1037.5 (290.62) | 1440.5 (593.01)
  A/Vietnam/1194/2004, min. 2 cytokines, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min. 2 cytokines, D42 | 4578.2 (848.69) | 5425.57 (2176.77) | 4917.67 (1787.62) | 3862.00 (1024.44) | 1024.5 (547.92) | 1492.6 (442.25)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D21 | 2516.33 (1390.64) | 5460.33 (3093.55) | 3606.00 (1871.46) | 3828.00 (1332.47) | 893 (298.4) | 1429.75 (603.52)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D42 | 4367.00 (858.47) | 5307.29 (2255.72) | 4863.50 (1767.69) | 3769.75 (980.19) | 1046.75 (550.36) | 1496.4 (416.88)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D21 | 2405.50 (1357.76) | 5345.00 (2828.98) | 3385.17 (1752.85) | 3708.75 (1542.48) | 925 (272.94) | 1412.5 (631.94)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D42 | 3981.40 (611.95) | 5008.14 (1938.05) | 4447.17 (1591.81) | 3461.25 (973.71) | 864 (428.27) | 1422.4 (432.38)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D21 | 1459.00 (947.19) | 2799.00 (2049.50) | 1636.33 (822.50) | 1741.50 (817.26) | 667.5 (144.96) | 951 (439.73)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D42 | 2570.60 (874.72) | 2573.71 (1258.22) | 2313.17 (956.59) | 1706.00 (298.05) | 667.5 (477.67) | 913.2 (262.45)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D21 | 1835.33 (1124.45) | 3822.67 (3294.28) | 2683.00 (1560.15) | 1995.50 (736.97) | 447.5 (258.09) | 890.75 (169.87)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D42 | 2813.40 (1327.05) | 4047.71 (2556.46) | 3670.00 (1922.75) | 2493.25 (1000.61) | 603 (590.71) | 733.8 (378.22)

28. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 8+ (CD8+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation
Description: as for outcome 27
Time Frame: Within 21 days of each primary vaccine dose: at Day 21 and at Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-cells per million cells
Arm/Group | H5N1 Adjuvanted Group - Lot 1 | H5N1 Adjuvanted Group - Lot 2 | H5N1 Adjuvanted Group - Lot 3 | H5N1 Adjuvanted Group - Lot 4 | H5N1 Un-Adjuvanted Group - Lot 1 | H5N1 Un-Adjuvanted Group - Lot 2
Number analyzed (Participants) | 6 | 7 | 6 | 4 | 4 | 5
T-cells per million cells
  A/Vietnam/1194/2004,min. 2 cytokines, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004,min. 2 cytokines, D21 | 166.0 (182.34) | 236.33 (177.38) | 76.67 (116) | 127 (122.34) | 289.5 (225.57) | 785.5 (1531.24)
  A/Vietnam/1194/2004, min. 2 cytokines, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min. 2 cytokines, D42 | 161 (128.26) | 176.43 (204.71) | 69.17 (67.19) | 32.5 (32.3) | 147 (125.63) | 172 (305.46)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D21 | 25.33 (30.73) | 1.00 (0) | 18.50 (20.74) | 1 (0) | 1 (0) | 78 (136.59)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, D42 | 15.20 (31.75) | 12.71 (30.99) | 13.50 (19.49) | 10.25 (11.06) | 1 (0) | 47.8 (33.69)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D21 | 144.33 (165.58) | 131.67 (70.81) | 66.17 (104.61) | 120.75 (153.51) | 198 (278.6) | 341.5 (663.12)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, D42 | 140.00 (148.92) | 108.71 (114.78) | 80.83 (73.51) | 30.00 (22.77) | 139 (103.58) | 138.6 (205.65)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D21 | 163.50 (187.70) | 245.33 (170.81) | 59.83 (89.57) | 104.75 (136.03) | 335 (229.1) | 765.25 (1510.55)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, D42 | 166.60 (131.04) | 161.29 (201.37) | 34.50 (43.63) | 23.75 (26.30) | 128.75 (138.81) | 159.8 (319.18)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D21: number analyzed (Participants) | 6 | 3 | 6 | 4 | 2 | 4
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D21 | 75.83 (135.65) | 175.33 (195.41) | 45.83 (74.25) | 95.25 (32.26) | 208.5 (12.02) | 804 (1485.55)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D42: number analyzed (Participants) | 5 | 7 | 6 | 4 | 4 | 5
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, D42 | 89.20 (64.10) | 164.14 (194.30) | 72.50 (100.04) | 29.75 (34.98) | 79.5 (127.03) | 110 (227.33)

29. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 4+ (CD4+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation
Description: as for outcome 27
Time Frame: as for outcome 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-cells per million T-cells
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 7 | 8
T-cells per million T-cells
  A/Vietnam/1194/2004, min. 2 cytokines, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min. 2 cytokines, M6 | 1773.0 (748.95) | 681.00 (243.30)
  A/Vietnam/1194/2004, min. 2 cytokines, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min. 2 cytokines, M6+21D | 7049.60 (3832.18) | 3898.00 (1133.03)
  A/Vietnam/1194/2004, min. 2 cytokines, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min. 2 cytokines, M6+42D |  | 4472.75 (2352.87)
  A/Vietnam/1194/2004, min. 2 cytokines, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min. 2 cytokines, M12 | 3197.29 (1428.81) | 2141.57 (617.49)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6 | 1720.00 (765.05) | 666 (187.51)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+21D | 6849.60 (3814.40) | 3885.60 (1116.51)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+42D |  | 4330.88 (2255.37)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12 | 3164.43 (1419.03) | 2148.57 (617.94)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6 | 921.00 (489.49) | 409.00 (227.75)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+21D | 3585.40 (2106.34) | 1665.60 (659.04)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+42D |  | 2332.25 (1640.24)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M12 | 1592.57 (781.64) | 1016.86 (509.21)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6 | 1653.33 (608.11) | 688.33 (212.18)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+21D | 6526.40 (3484.66) | 3674.00 (1062.72)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+42D |  | 4177.25 (2092.28)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12 | 3043.86 (1386.80) | 2098.86 (558.63)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6 | 1443.00 (554.28) | 538.33 (224.38)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+21D | 5544.20 (3219.20) | 2671.00 (863.72)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+42D |  | 3296.25 (2060.05)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12 | 2501.43 (1190.18) | 1649.14 (504.41)

30. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 8+ (CD8+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation
Description: The analyzed cytokines were CD40 Ligand (CD40L), Interleukin 2 (IL-2), Tumor Necrosis Factor-α (TNF-α) and Interferon-γ (IFN-γ). The stimulating antigen used was A/Vietnam/1194/2004.
Time Frame: as for outcome 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-cells per million T-cells
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 7 | 8
T-cells per million T-cells
  A/Vietnam/1194/2004, min. 2 cytokines, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min. 2 cytokines, M6 | 55.00 (49.76) | 306.00 (363.19)
  A/Vietnam/1194/2004, min. 2 cytokines, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min. 2 cytokines, M6+21D | 50.00 (47.94) | 62.60 (47.45)
  A/Vietnam/1194/2004, min. 2 cytokines, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min. 2 cytokines, M6+42D |  | 257.63 (484.86)
  A/Vietnam/1194/2004, min. 2 cytokines, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min. 2 cytokines, M12 | 50.86 (75.46) | 232.00 (383.34)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6 | 3.67 (4.62) | 5.33 (7.51)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+21D | 23.80 (24.65) | 31.20 (52.39)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6+42D |  | 5.38 (10.85)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12 | 12.29 (12.11) | 4.71 (9.83)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6 | 44 (37.24) | 331.33 (407.67)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+21D | 36 (30.74) | 50.60 (40.5)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6+42D |  | 257 (485.24)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M12 | 53 (83.7) | 211.71 (375.25)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6 | 22.67 (33.29) | 162.00 (229.00)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+21D | 39.40 (38.00) | 36.60 (33.08)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6+42D |  | 147.88 (246.47)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12 | 38.00 (52.50) | 133.14 (168.94)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6: number analyzed (Participants) | 3 | 3
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6 | 58.67 (58.52) | 290 (335.72)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+21D: number analyzed (Participants) | 5 | 5
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+21D | 24.6 (23.56) | 219.88 (443.7)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+42D: number analyzed (Participants) | 0 | 8
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6+42D |  | 219.88 (443.7)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12: number analyzed (Participants) | 7 | 7
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12 | 34 (63.9) | 204.43 (376.77)

31. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 4+ (CD4+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation for Subjects Not Boosted at Month 6
Description: as for outcome 27
Time Frame: At Month 6 and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-cells per million T-cells
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 30
T-cells per million T-cells
  A/Vietnam/1194/2004, min. 2 cytokines, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min. 2 cytokines, M6 | 2529.54 (1063.65)
  A/Vietnam/1194/2004, min. 2 cytokines, M12 | 2098.17 (1287.49)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6 | 2407.31 (1009.26)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12 | 2004.27 (1193.53)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6 | 1387.38 (840.81)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M12 | 1184.07 (992.44)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6 | 2341.15 (936.20)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12 | 1912.60 (1130.58)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6 | 1960.62 (891.12)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12 | 1599.20 (945.88)

32. Secondary Outcome: Frequency of Influenza-specific Cluster of Differentiation 8+ (CD8+) T Cells Expressing at Least 2 Markers Among the Analyzed Cytokines Upon in Vitro Stimulation for Subjects Not Boosted at Month 6
Description: as for outcome 27
Time Frame: At Month 6 and at Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-cells per million T-cells
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 30
T-cells per million T-cells
  A/Vietnam/1194/2004, min. 2 cytokines, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min. 2 cytokines, M6 | 82.69 (166.59)
  A/Vietnam/1194/2004, min. 2 cytokines, M12 | 106.13 (173.19)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M6 | 9.62 (13.90)
  A/Vietnam/1194/2004, min. CD40L+1 cytokine, M12 | 4.53 (8.18)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M6 | 67.23 (145.99)
  A/Vietnam/1194/2004, min.IFN-γ+1 cytokine, M12 | 102.93 (161.31)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M6 | 66.00 (117.35)
  A/Vietnam/1194/2004, min.IL-2+1 cytokine, M12 | 70.90 (128.03)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6: number analyzed (Participants) | 13
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M6 | 59.08 (111.73)
  A/Vietnam/1194/2004, min.TNF-α+1 cytokine, M12 | 89.30 (140.96)

33. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-days (Days 0-6) post-primary vaccination period following each dose and overall
Population: The analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects who had completed their symptom sheet for the considered timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 954 | 245
Participants
  Any Ecchymosis, Dose 1 | 8 | 0
  Grade 3 Ecchymosis, Dose 1 | 0 | 0
  Any Induration, Dose 1 | 54 | 0
  Grade 3 Induration, Dose 1 | 0 | 0
  Any Pain, Dose 1 | 779 | 44
  Grade 3 Pain, Dose 1 | 31 | 0
  Any Redness, Dose 1 | 36 | 0
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 84 | 0
  Grade 3 Swelling, Dose 1 | 1 | 0
  Any Ecchymosis, Dose 2: number analyzed (Participants) | 944 | 245
  Any Ecchymosis, Dose 2 | 3 | 0
  Grade 3 Ecchymosis, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Ecchymosis, Dose 2 | 0 | 0
  Any Induration, Dose 2: number analyzed (Participants) | 944 | 245
  Any Induration, Dose 2 | 38 | 0
  Grade 3 Induration, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Induration, Dose 2 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 944 | 245
  Any Pain, Dose 2 | 674 | 38
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Pain, Dose 2 | 21 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 944 | 245
  Any Redness, Dose 2 | 33 | 1
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 944 | 245
  Any Swelling, Dose 2 | 70 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Ecchymosis, Across doses | 10 | 0
  Grade 3 Ecchymosis, Across doses | 0 | 0
  Any Induration, Across doses | 76 | 0
  Grade 3 Induration, Across doses | 0 | 0
  Any Pain, Across doses | 830 | 62
  Grade 3 Pain, Across doses | 49 | 0
  Any Redness, Across doses | 64 | 1
  Grade 3 Redness, Across doses | 1 | 0
  Any Swelling, Across doses | 114 | 0
  Grade 3 Swelling, Across doses | 1 | 0

34. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-days (Days 0-6) post-primary vaccination period following each dose and overall
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 954 | 245
Participants
  Any Arthralgia, Dose 1 | 118 | 16
  Grade 3 Arthralgia, Dose 1 | 5 | 0
  Related Arthralgia, Dose 1 | 109 | 14
  Any Fatigue , Dose 1 | 411 | 69
  Grade 3 Fatigue , Dose 1 | 18 | 0
  Related Fatigue , Dose 1 | 395 | 65
  Any Fever, Dose 1 | 21 | 1
  Grade 3 Fever, Dose 1 | 5 | 0
  Related Fever, Dose 1 | 20 | 1
  Any Headache, Dose 1 | 238 | 35
  Grade 3 Headache, Dose 1 | 13 | 0
  Related Headache, Dose 1 | 215 | 29
  Any Myalgia, Dose 1 | 478 | 48
  Grade 3 Myalgia, Dose 1 | 14 | 0
  Related Myalgia, Dose 1 | 462 | 43
  Any Shivering, Dose 1 | 44 | 3
  Grade 3 Shivering, Dose 1 | 2 | 0
  Related Shivering, Dose 1 | 42 | 2
  Any Sweating, Dose 1 | 86 | 19
  Grade 3 Sweating, Dose 1 | 0 | 0
  Related Sweating, Dose 1 | 78 | 17
  Any Arthralgia, Dose 2: number analyzed (Participants) | 944 | 245
  Any Arthralgia, Dose 2 | 147 | 14
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Arthralgia, Dose 2 | 4 | 1
  Related Arthralgia, Dose 2: number analyzed (Participants) | 944 | 245
  Related Arthralgia, Dose 2 | 147 | 13
  Any Fatigue , Dose 2: number analyzed (Participants) | 944 | 245
  Any Fatigue , Dose 2 | 435 | 53
  Grade 3 Fatigue , Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Fatigue , Dose 2 | 26 | 2
  Related Fatigue , Dose 2: number analyzed (Participants) | 944 | 245
  Related Fatigue , Dose 2 | 432 | 52
  Any Fever, Dose 2: number analyzed (Participants) | 944 | 245
  Any Fever, Dose 2 | 27 | 3
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Fever, Dose 2 | 3 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 944 | 245
  Related Fever, Dose 2 | 27 | 3
  Any Headache, Dose 2: number analyzed (Participants) | 944 | 245
  Any Headache, Dose 2 | 269 | 29
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Headache, Dose 2 | 16 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 944 | 245
  Related Headache, Dose 2 | 265 | 27
  Any Myalgia, Dose 2: number analyzed (Participants) | 944 | 245
  Any Myalgia, Dose 2 | 429 | 34
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Myalgia, Dose 2 | 17 | 1
  Related Myalgia, Dose 2: number analyzed (Participants) | 944 | 245
  Related Myalgia, Dose 2 | 427 | 34
  Any Shivering, Dose 2: number analyzed (Participants) | 944 | 245
  Any Shivering, Dose 2 | 75 | 4
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Shivering, Dose 2 | 4 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 944 | 245
  Related Shivering, Dose 2 | 74 | 4
  Any Sweating, Dose 2: number analyzed (Participants) | 944 | 245
  Any Sweating, Dose 2 | 90 | 13
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 944 | 245
  Grade 3 Sweating, Dose 2 | 4 | 2
  Related Sweating, Dose 2: number analyzed (Participants) | 944 | 245
  Related Sweating, Dose 2 | 87 | 13
  Any Arthralgia, Across doses | 212 | 24
  Grade 3 Arthralgia, Across doses | 8 | 1
  Related Arthralgia, Across doses | 206 | 22
  Any Fatigue , Across doses | 559 | 91
  Grade 3 Fatigue , Across doses | 38 | 2
  Related Fatigue , Across doses | 550 | 88
  Any Fever, Across doses | 45 | 4
  Grade 3 Fever, Across doses | 8 | 1
  Related Fever, Across doses | 44 | 4
  Any Headache, Across doses | 380 | 52
  Grade 3 Headache, Across doses | 26 | 1
  Related Headache, Across doses | 367 | 47
  Any Myalgia, Across doses | 610 | 65
  Grade 3 Myalgia, Across doses | 29 | 1
  Related Myalgia, Across doses | 599 | 61
  Any Shivering, Across doses | 105 | 7
  Grade 3 Shivering, Across doses | 6 | 1
  Related Shivering, Across doses | 103 | 6
  Any Sweating, Across doses | 143 | 25
  Grade 3 Sweating, Across doses | 4 | 2
  Related Sweating, Across doses | 135 | 24

35. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Booster Phase
Description: as for outcome 33
Time Frame: During the 7-days (Days 0-6) post-booster vaccination period
Population: The analysis was performed on the Booster Total Vaccinated Cohort, including all vaccinated subjects who were boosted at Month 6 and who had completed their symptom sheet for the considered timepoint. Considering subjects from H5N1 Adjuvanted Group only received one single booster dose, data are reported only for booster dose 1 for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 265 | 235
Participants
  Any Ecchymosis, Booster dose 1 | 2 | 1
  Grade 3 Ecchymosis, Booster dose 1 | 0 | 0
  Any Induration, Booster dose 1 | 21 | 14
  Grade 3 Induration, Booster dose 1 | 0 | 1
  Any Pain, Booster dose 1 | 214 | 187
  Grade 3 Pain, Booster dose 1 | 14 | 11
  Any Redness, Booster dose 1 | 16 | 7
  Grade 3 Redness, Booster dose 1 | 0 | 0
  Any Swelling, Booster dose 1 | 36 | 24
  Grade 3 Swelling, Booster dose 1 | 0 | 0
  Any Ecchymosis, Booster dose 2: number analyzed (Participants) | 265 | 234
  Any Ecchymosis, Booster dose 2 | 0 | 2
  Grade 3 Ecchymosis, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Ecchymosis, Booster dose 2 |  | 0
  Any Induration, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Induration, Booster dose 2 |  | 14
  Grade 3 Induration, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Induration, Booster dose 2 |  | 0
  Any Pain, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Pain, Booster dose 2 |  | 159
  Grade 3 Pain, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Pain, Booster dose 2 |  | 8
  Any Redness, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Redness, Booster dose 2 |  | 15
  Grade 3 Redness, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Redness, Booster dose 2 |  | 0
  Any Swelling, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Swelling, Booster dose 2 |  | 22
  Grade 3 Swelling, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Swelling, Booster dose 2 |  | 0
  Any Ecchymosis, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Ecchymosis, Across booster doses |  | 2
  Grade 3 Ecchymosis, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Ecchymosis, Across booster doses |  | 0
  Any Induration, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Induration, Across booster doses |  | 21
  Grade 3 Induration, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Induration, Across booster doses |  | 1
  Any Pain, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Pain, Across booster doses |  | 198
  Grade 3 Pain, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Pain, Across booster doses |  | 17
  Any Redness, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Redness, Across booster doses |  | 16
  Grade 3 Redness, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Redness, Across booster doses |  | 0
  Any Swelling, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Swelling, Across booster doses |  | 33
  Grade 3 Swelling, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Swelling, Across booster doses |  | 0

36. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms - Booster Phase
Description: as for outcome 34
Time Frame: During the 7-days (Days 0-6) post-booster vaccination period
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 265 | 235
Participants
  Any Arthralgia, Booster dose 1 | 57 | 33
  Grade 3 Arthralgia, Booster dose 1 | 4 | 1
  Related Arthralgia, Booster dose 1 | 57 | 32
  Any Fatigue , Booster dose 1 | 165 | 96
  Grade 3 Fatigue , Booster dose 1 | 15 | 3
  Related Fatigue , Booster dose 1 | 164 | 95
  Any Fever, Booster dose 1 | 16 | 7
  Grade 3 Fever, Booster dose 1 | 3 | 0
  Related Fever, Booster dose 1 | 16 | 7
  Any Headache, Booster dose 1 | 120 | 66
  Grade 3 Headache, Booster dose 1 | 8 | 1
  Related Headache, Booster dose 1 | 117 | 65
  Any Myalgia, Booster dose 1 | 169 | 126
  Grade 3 Myalgia, Booster dose 1 | 15 | 4
  Related Myalgia, Booster dose 1 | 168 | 126
  Any Shivering, Booster dose 1 | 47 | 18
  Grade 3 Shivering, Booster dose 1 | 5 | 0
  Related Shivering, Booster dose 1 | 47 | 18
  Any Sweating, Booster dose 1 | 25 | 15
  Grade 3 Sweating, Booster dose 1 | 0 | 0
  Related Sweating, Booster dose 1 | 23 | 15
  Any Arthralgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Arthralgia, Booster dose 2 |  | 38
  Grade 3 Arthralgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Arthralgia, Booster dose 2 |  | 3
  Related Arthralgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Arthralgia, Booster dose 2 |  | 37
  Any Fatigue , Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Fatigue , Booster dose 2 |  | 95
  Grade 3 Fatigue , Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Fatigue , Booster dose 2 |  | 4
  Related Fatigue , Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Fatigue , Booster dose 2 |  | 94
  Any Fever, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Fever, Booster dose 2 |  | 9
  Grade 3 Fever, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Fever, Booster dose 2 |  | 1
  Related Fever, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Fever, Booster dose 2 |  | 9
  Any Headache, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Headache, Booster dose 2 |  | 69
  Grade 3 Headache, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Headache, Booster dose 2 |  | 3
  Related Headache, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Headache, Booster dose 2 |  | 68
  Any Myalgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Myalgia, Booster dose 2 |  | 101
  Grade 3 Myalgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Myalgia, Booster dose 2 |  | 5
  Related Myalgia, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Myalgia, Booster dose 2 |  | 100
  Any Shivering, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Shivering, Booster dose 2 |  | 30
  Grade 3 Shivering, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Shivering, Booster dose 2 |  | 2
  Related Shivering, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Shivering, Booster dose 2 |  | 29
  Any Sweating, Booster dose 2: number analyzed (Participants) | 0 | 234
  Any Sweating, Booster dose 2 |  | 21
  Grade 3 Sweating, Booster dose 2: number analyzed (Participants) | 0 | 234
  Grade 3 Sweating, Booster dose 2 |  | 1
  Related Sweating, Booster dose 2: number analyzed (Participants) | 0 | 234
  Related Sweating, Booster dose 2 |  | 21
  Any Arthralgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Arthralgia, Across booster doses |  | 54
  Grade 3 Arthralgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Arthralgia, Across booster doses |  | 4
  Related Arthralgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Arthralgia, Across booster doses |  | 52
  Any Fatigue , Across booster doses: number analyzed (Participants) | 0 | 235
  Any Fatigue , Across booster doses |  | 121
  Grade 3 Fatigue , Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Fatigue , Across booster doses |  | 6
  Related Fatigue , Across booster doses: number analyzed (Participants) | 0 | 235
  Related Fatigue , Across booster doses |  | 119
  Any Fever, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Fever, Across booster doses |  | 14
  Grade 3 Fever, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Fever, Across booster doses |  | 1
  Related Fever, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Fever, Across booster doses |  | 14
  Any Headache, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Headache, Across booster doses |  | 97
  Grade 3 Headache, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Headache, Across booster doses |  | 3
  Related Headache, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Headache, Across booster doses |  | 96
  Any Myalgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Myalgia, Across booster doses |  | 141
  Grade 3 Myalgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Myalgia, Across booster doses |  | 9
  Related Myalgia, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Myalgia, Across booster doses |  | 141
  Any Shivering, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Shivering, Across booster doses |  | 38
  Grade 3 Shivering, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Shivering, Across booster doses |  | 2
  Related Shivering, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Shivering, Across booster doses |  | 37
  Any Sweating, Across booster doses: number analyzed (Participants) | 0 | 235
  Any Sweating, Across booster doses |  | 28
  Grade 3 Sweating, Across booster doses: number analyzed (Participants) | 0 | 235
  Grade 3 Sweating, Across booster doses |  | 1
  Related Sweating, Across booster doses: number analyzed (Participants) | 0 | 235
  Related Sweating, Across booster doses |  | 28

37. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the primary phase (from Day 0 to Month 6)
Population: The analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects for whom data were available for the considered timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 961 | 245
Participants | 308 | 75

38. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 37
Time Frame: During the booster phase (from Month 6 to Month 12)
Population: The analysis was performed on the Booster Total Vaccinated Cohort, including all vaccinated subjects who were boosted at Month 6 and for whom data were available for the considered timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 265 | 236
Participants | 65 | 54

39. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the primary phase (from Day 0 to Month 6)
Population: The analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects for whom were available for the considered timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 961 | 245
Participants | 7 | 0

40. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: as for outcome 39
Time Frame: During the booster phase (from Month 6 to Month 12)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
Number analyzed (Participants) | 265 | 236
Participants | 3 | 5

41. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) for Subjects Not Boosted at Month 6
Description: This group consists of the remaining subjects from the GSK1562902A Pooled Group who received a single dose of H5N1 vaccine at Month 12 or 36.
Time Frame: From Month 6 to Month 12
Population: The analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects who were not boosted at Month 6 (Non-Boosted sub-cohort) and for whom data were available for the considered timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Adjuvanted Group
Number analyzed (Participants) | 672
Participants | 15

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7-day post-vaccination period (Days 0-6), Unsolicited AEs up to 21 days (Day 0-20) after the first vaccination and 30 days (Day 0-29) after the second vaccination, SAEs during the entire study period (Day 0 - Month 12).
Arm/Group | H5N1 Adjuvanted Group | H5N1 Un-adjuvanted Group
All-Cause Mortality (participants affected / at risk) | 1/961 | 0/245
Serious Adverse Events (participants affected / at risk) | 25/961 | 5/245
Other Adverse Events (participants affected / at risk) | 904/961 | 159/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H5N1 Adjuvanted Group (N=961) | H5N1 Un-adjuvanted Group (N=245)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Accidental death (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 3 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H5N1 Adjuvanted Group (N=961) | H5N1 Un-adjuvanted Group (N=245)
Chills (General disorders) | 105 (119) | 7 (7)
Fatigue (General disorders) | 559 (846) | 91 (122)
Induration (General disorders) | 246 (334) | 11 (11)
Injection site erythema (General disorders) | 321 (456) | 48 (67)
Injection site pain (General disorders) | 830 (1453) | 62 (82)
Injection site swelling (General disorders) | 365 (519) | 23 (31)
Pyrexia (General disorders) | 185 (213) | 21 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 214 (268) | 24 (30)
Myalgia (Musculoskeletal and connective tissue disorders) | 610 (909) | 65 (83)
Headache (Nervous system disorders) | 389 (527) | 59 (75)
Ecchymosis (Skin and subcutaneous tissue disorders) | 68 (77) | 10 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 143 (176) | 25 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.